CLINICAL TRIAL: NCT04580329
Title: The Effect of Neuromuscular Electrical Stimulation (NMES) on the Renal Function and Renal Blood Flow for Patients With Pregnancy Related- Acute Kidney Injury
Brief Title: The Effect of Neuromuscular Electrical Stimulation (NMES) on the Renal Function and Renal Blood Flow
Acronym: NMES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ahmed talaat ahmed aly (Other)
Responsible Party: Sponsor-Investigator, Ahmed talaat ahmed aly, clinical professor, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NMES
Record Dates: First submitted 2020-09-30; First posted 2020-10-08 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Renal Injury
Keywords: neuromuscular electrical stimulation; renal function; renal blood flow; Acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMES group (Experimental)
  Interventions: Procedure: neuromuscular electrical stimulation (NMES) in addition to routine hospital care
- control group (Experimental)
  Interventions: Procedure: routine hospital care without NMES

INTERVENTIONS:
Procedure: neuromuscular electrical stimulation (NMES) in addition to routine hospital care — Patients in the NMES group will receive NMES sessions as the electrodes will be placed around the bilateral femoral quadriceps muscles and at the site of renal arteries.
  NMES(>100 Hz, 50-80 μ sec) will be performed for 55 min including 5 minutes for warm up and 5 minutes for recovery .
  The intensity of electrical stimulation will be adjusted to suit the comfort level of each individual patient without producing discomfort or pain.
  Arms: NMES group
Procedure: routine hospital care without NMES — routine hospital care include all the routine intervention done for post partum women with AKI including fluid resuscitation, diuretics, hemodialysis
  Arms: control group

SUMMARY:
A randomized prospective controlled study aims to evaluate the effect of neuromuscular electrical stimulation on the renal function and renal blood flow of post partum women with acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or old and hemodynamically stable.
* Post-partum women who developed AKI.

Exclusion Criteria:

* Pregnant women .
* Patients who required any emergency or elective surgery during the study; those who presented acute heart or lung disease, skin rashes, tumors, infections, diabetes mellitus or hypoesthesia in the region that the neuromuscular electrical stimulation would be applied.
* Patients with a Pacemaker.
* Epileptic Patients.
* Patients with recent effects of stroke (less than 3 months).
* Uncontrolled hypertension (systolic blood pressure > 230 mm Hg and diastolic blood pressure > 120 mm Hg).

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
renal function change | for 7 days
  serum creatinine level will be assessed and it will show improvement
renal blood flow change | for 7 days
  urine output will be assessed and it will show improvement

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed T Ahmed, A professor, Principal Investigator — Assiut University
Locations (1):
- Ahmed Talaat Ahmed, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No